CLINICAL TRIAL: NCT01270256
Title: Evaluation of NasoNeb™ Delivery of an Intranasal Steroid in the Treatment of Perennial Allergic Rhinitis
Brief Title: NasoNeb Delivery of an Intranasal Steroid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: MedInvent, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-660-B
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Perennial Allergic Rhinitis
Keywords: allergy
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Hypersensitivity | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide (Active Comparator): Pulmicort Respules at a dose of 0.25 mg. delivered intranasally via NasoNeb nebulizer once daily
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Placebo delivered intranasally via NasoNeb nebulizer once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — Pulmicort Respules at a dose of 0.25 mg. delivered intranasally via NasoNeb nebulizer once daily
  Arms: Budesonide
Drug: Placebo — Placebo delivered intranasally via NasoNeb nebulizer once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if a nasal steroid drug delivered to the nose with the NasoNeb™ inhaler improves the symptoms of people with perennial allergic rhinitis (year round allergy symptoms).

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 55 years of age.
2. History of perennial allergic rhinitis.
3. Positive skin test to dust mite, dog, cat or indoor mold antigen.
4. And a combined nasal AM and PM score of ≥4 for nasal congestion in the day preceding entry and total nasal symptom score greater than 8.

Exclusion Criteria

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Subjects treated with systemic steroids during the previous 30 days.
4. Subjects treated with topical (inhaled, intranasal or intraocular) steroids, Nasalcrom or Opticrom during the previous 30 days.
5. Subjects treated with oral antihistamine/decongestants during the previous seven days.
6. Subjects treated with topical (intranasal or intraocular) antihistamine/decongestants during the previous 3 days.
7. Subjects treated with immunotherapy and are escalating their dose.
8. Subjects on chronic anti-asthma medications.
9. Subjects with polyps in the nose or a significantly displaced septum.
10. Upper respiratory infection within 14 days prior to study start.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Brown K, Lane J, Silva MP, DeTineo M, Naclerio RM, Baroody FM. A pilot study of the effects of intranasal budesonide delivered by NasoNeb(R) on patients with perennial allergic rhinitis. Int Forum Allergy Rhinol. 2014 Jan;4(1):43-8. doi: 10.1002/alr.21239. PMID 24574125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Budesonide | Placebo
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 33.3 [18 to 55] | 32.3 [18 to 52] | 32.8 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Nasal Peak Inspiratory Flow (NPIF)
Description: NPIF was measured objectively in liters per minute with an In-Check Peak & Inspiratory Flow Meter (Ferraris Medical Inc, Orchard Park, NY). Subjects obtained 3 readings every morning and every evening and the greatest of the 3 measures were recorded. Total daily NPIF was calculated by adding the morning and evening values each day and the average of the change from baseline in NPIF for all days of was calculated
Time Frame: Baseline and 26 days
Measure: Median (Standard Error); unit: liters/min
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 20 | 20
liters/min | 36.41 (8.9) | 18.71 (8.37)

ADVERSE EVENTS:
Arm/Group | Budesonide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes